CLINICAL TRIAL: NCT05545085
Title: Thoracoscopic Laser Speckle Contrast Imaging for the Demarcation of Lung Segments
Brief Title: Thoracoscopic Laser Speckle Contrast Imaging for Segment Resections
Acronym: PORTION-I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University of Groningen (Other); LIMIS Development (Unknown)
Responsible Party: Principal Investigator, E.C. Boerma, Dr., Frisius Medisch Centrum
Other Study IDs: NL82338.099.22
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All included patients meeting the eligibility criteria and scheduled to undergo a lobectomy in the Medical Centre Leeuwarden.
  Interventions: Device: Laser Speckle Contrast Imaging using the PerfusiX-Imaging Device

INTERVENTIONS:
Device: Laser Speckle Contrast Imaging using the PerfusiX-Imaging Device — Patient will undergo the standard of care lobectomy for pulmonary cancer. In addition, peroperative imaging using the Laser Speckle Contrast Imaging device will be performed.

SUMMARY:
Rationale Lung cancer remains to be the leading cause of cancer-related deaths worldwide1. The current standard-of-care for small lung cancer is a total lobectomy. Albeit effective with respect to the radical excision of the tumour, the substantial loss in lung tissue may be clinically relevant, especially in combination with frequently co-existing lung diseases. Thoracoscopic segmentectomy is a combination of adequate oncological resection with lung-tissue-sparing properties and is being increasingly used because of its several advantages compared with lobar resections. By defining the segment that has to be excised pre-operatively, the key to successful pulmonary segmentectomy is to subsequently intraoperatively recognize the intersegmental planes correctly. The conventional and most common method uses a ventilation method (inflation/deflation technique). With the increasing availability of endoscopic imaging systems, indocyanine green (ICG) fluorescence imaging is a more advanced method to determine intersegmental planes. The major limitation is the use of an exogenous contrast agent. After injection, the ICG only has very limited "imaging time window" (minutes) in which the images can be used to determine the intersegmental planes. Furthermore, the use of dye limits repeatability of measurements due to rest ICG, the extra operating room time required for the injection, wash-in and wash-out of the dye as well as change of camera settings. These limitations leave room for new technologies and improvements. The investigators hypothesized that an endoscopic laser speckle imaging device could overcome the limitations of ICG-fluorescence imaging and could thus be a very useful addition in intersegmental plane detection. PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands) is such an endoscopic laser speckle contrast imager that has been developed in the Medical Centre Leeuwarden since 2014. LSCI has never been used to identify intersegmental planes, however, based on the similarities between LSCI and ICG-fluorescence, this novel imaging approach is thought to be effective and potentially could be used as a standard-of-care.

Objectives In this trial the investigators will study the utility of PerfusiX-Imaging for the identification of intersegmental planes during thoracoscopic segmentectomy.

Study design The current study is a prospective, observational single-centre study in the Medical Center Leeuwarden.

Study population A total of 10 patients undergoing an upper left or right lobectomy. Patient related study procedures All patients will undergo the standard-of-care program which includes perfusion assessment by ICG-fluorescence imaging. In addition to this standard-of-care, 2D-perfusion maps will be generated from images taken with PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands). Not related to the patient, the PerfusiX-Imaging images will be shown to the surgeon postoperatively and peroperative questionnaires will be filled regarding the standard-of-care perfusion assessment.

Study parameters/endpoints Due to the explorative character of this study, there is no formal hierarchy in the respective endpoints of this study. In this, all endpoints will add to the overall assessment of the feasibility of the PerfusiX-imaging derived visual feedback for detecting interlobar and intersegmental planes in lung tissue. The investigators will register whether it was possible to detect the intersegmental plane. Subsequently, compare the difference in location of both the interlobar and intersegmental planes as derived from visual feedback from the PerfusiX-imaging system is compared, with images derived from ICG imaging and the surgical eye. During the procedure, the time needed to generate and acquire the visual feedback from the PerfusiX-imaging system will be determined. The investigators will also determine the interpretability of the visual feedback from the PerfusiX-imaging system by users (surgeons). In addition, the investigators will determine Laser Speckle Perfusion Unit (LSPU) cut-off values of PerfusiX-imaging in lung tissue with the best sensitivity and specificity for the indication of level of tissue perfusion.

Burden, risk and benefit to participation Burden Not applicable. Risks Not applicable. Benefit Not applicable.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE 1.1 General introduction Despite recent major improvements in diagnosis, staging and treatment, lung cancer remains to be the leading cause of cancer-related deaths worldwide. Since the demonstration of superiority over sublobar lung resection, the current standard-of-care for small lung cancer is a lobectomy. In a lobectomy, one of the three (right lung) or two (left lung) lobes is excised. Albeit effective with respect to the radical excision of the tumour, the substantial loss in lung tissue may be clinically relevant, especially in combination with frequently co-existing lung diseases. This is made possible due to high resolution medical imaging (computed tomography) that enables surgeons to precisely locate small tumors. This paved the way for segmentectomy. Thoracoscopic segmentectomy is a combination of adequate oncological resection with lung-tissue-sparing properties and is being increasingly used because of its several advantages compared with lobar resections. Local recurrences after surgical resection are correlated to the length of the safety margins. These margins are defined by guidelines (2 cm for tumours >2 cm or a margin that is at least as large as the tumour diameter for smaller lesions). By defining the segment that has to be excised pre-operatively, the key to successful pulmonary segmentectomy is to subsequently intraoperatively recognize the intersegmental planes correctly. Although the intersegmental plane is regulated by intersegmental veins, it would be impossible to detect and follow these veins in the distal lung parenchyma, therefore, it is mandatory to identify the intersegmental plane before dividing the lung parenchyma.

1.2 Intersegmental plane detection methods The conventional and most common way to intraoperatively identify the intersegmental plane uses a conventional ventilation method (inflation/deflation technique). The targeted segment may be isolated from the rest of the lobe by selectively inflating the residual segments leaving the target segment atelectatic or, on the contrary, may be selectively inflated leaving the rest of the lobe atelectatic. A limitation of this method is the limited space to manoeuvre during video-assisted surgery.

More recently, optical imaging-based image guided surgery approaches are being developed to intraoperatively identify the intersegmental planes. With the increasing availability of endoscopic fluorescence imaging systems comes the popularity of fluorescence imaging throughout all surgical fields. This led to the development of methylene blue for intersegmental plane identification. However, the most common approach is the use of indocyanine green (ICG) fluorescence imaging. ICG-fluorescence imaging is based on the excitation of ICG, which is an exogenous contrast agent that is intravenously injected. The ICG binds to blood proteins that starts to circulate and gets excreted via the liver.

The ICG enables the surgeon to clearly identify the intersegmental planes after ligation of the main feeding artery. This method shows great potential but comes with limitations. The major limitation is the use of an exogenous contrast agent. After injection, the ICG only has very limited "imaging time window" (minutes) in which the images can be used to determine the intersegmental planes. In practice, this means that the surgeon quickly marks the intersegmental plane using an energy device. In an ideal situation the surgeon has as long as required for this action. Furthermore, the use of dye limits repeatability of measurements due to rest ICG, the extra operating room time required for the injection, wash-in and wash-out of the dye as well as change of camera settings.

1.3 Laser speckle contrast imaging for intersegmental plane detection ICG fluorescence imaging is a perfusion imaging technique that can help identify the intersegmental plane based on a perfusion difference that is created by ligation of the main feeding artery of the segment of interest. After ligation, ICG is infused. The distribution of ICG is visualized on the monitor, using a near-infrared camerasystem. The isolated segment will not exhibit any fluorescent signal and will therewith be identifiable using ICG. Laser speckle contrast imaging (LSCI) is a perfusion imaging technique that seems to have similar use cases as ICG with the added advantage of not using exogenous contrast. LSCI. The first biomedical application of LSCI was reported in the 1981 by Fercher and Briers. The proposed technique from Fercher and Briers was non-real-time and had its practical limitations due to the use of non-digital systems which impeded the clinical use. The first real speed increase to quasi real-time image acquisition and processing happened in the nineties with the introduction of digital photography. Generally, the components required are a low-powered laser diode, a diffuser, a digital camera and processing software.

The investigators hypothesized that an endoscopic laser speckle imaging device could overcome the limitations of ICG-fluorescence imaging and could thus be a very useful addition in intersegmental plane detection. PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands) is such an endoscopic laser speckle contrast imager that has been developed in the Medical Centre Leeuwarden since 2014. LSCI has never been used to identify intersegmental planes, however, based on the similarities between LSCI and ICG-fluorescence and their capability to visualize differences in tissue perfusion,, this novel imaging approach is thought to be effective and potentially could be used as a standard-of-care.

1.4 The basic principle of laser speckle contrast imaging Speckle patterns are the random interference patterns that arise when coherent light is backscattered by a scattering medium such as biological tissue. The slightly different optical pathlengths cause the waves to reach the observer at random mutual phases, resulting in bright and dark spots respectively. The speckle image is built up of static and dynamic speckles. Static speckles are speckles that do not change over time whereas dynamic speckles do change over time due to the optical Doppler effect. The dynamic speckles contain information about movement of the object, or motion of particles within the object.

In order to be able to detect a change in the speckle pattern, the exposure time of the camera must be of the order of the speckle decorrelation time, causing a blurring of the recorded speckle pattern. It is this blurring that is used to calculate the speckle contrast K using the following formula:

K=σ/(<I>) Where σ is the standard deviation of the intensity I over the mean intensity <I> calculated over a window in space or time. Spatial contrast uses an area of multiple pixels in one frame as can be seen in the bottom left corner of Figure 4. A window size of 5 x 5 or 7 x 7 pixels has been suggested for optimal results10. As spatial contrast decreases the spatial resolution, however, this method does have a high temporal resolution. Temporal LSCI uses the same pixel in multiple frames to calculate the contrast in a time window. Temporal contrast has a high spatial resolution and low temporal resolution. For spatial contrast this is vice versa and hence, it can be beneficial if combined into a so-called spatio-temporal contrast. The choice of resolution should be based on the need for a high temporal or spatial resolution.

If the exposure time of the detector is shorter than the intensity fluctuation time of the speckles, the standard deviation σ is equal to the mean intensity <I> which theoretically results in a contrast value of K=1. If there is movement present and the exposure time of the detector is of the order of, or longer than the fluctuation time, the picture will be blurred meaning that the standard deviation σ will be small compared to the mean intensity <I> which results in a loss of contrast, hence 0≥K<1. Other names for the same principle as LSCI are laser speckle imaging (LSI), laser speckle perfusion imaging (LSPI) and laser speckle contrast analysis (LASCA) as it was named by the first users.

1.5 Rationale for the PORTION-I study The investigators hypothesize that PerfusiX-Imaging can help improve intersegmental plane identification during thoracoscopic segmentectomy. The current intraoperative identification of intersegmental during segmental resections is based on subjective clinical indicators, i.e., the surgeon's eye and ICG-fluorescence imaging. ICG-fluorescence imaging is deemed a substantial improvement over solely the surgeons' eye, however, this approach comes with several limitations. The most important is the short effective imaging period which means that the surgeon only has a very limited amount of time to mark the intersegmental planes. Moreover, by using PerfusiX-Imaging, the surgeon does not have to deal with a short effective imaging period. This enables real-time identification of the segment, without the need of marking the planes with an energy device. In this prospective, observational feasibility study, the investigators aim to determine whether PerfusiX-Imaging is capable of successfully identifying lung segments. As there are no segmental resections performed in the Medical Centre Leeuwarden at this moment, the investigators will image the interlobar plane during an upper left or right lobectomy in 10 patients. Also, the investigators will image the sublobar segment in these patients during preparation for the lobectomy.

3. STUDY DESIGN The current study is a prospective, observational single-centre study in the Medical Center Leeuwarden. A total of 10 patients undergoing an upper left or upper right lobectomy will be included (see section 4 'Study population'). APatients will - after written informed consent - undergo the regular standard-of-care program. In addition to this standard-of-care, 2D-perfusion maps will be generated from images taken with PerfusiX-Imaging (LIMIS Development BV, Leeuwarden, The Netherlands) in combination with a standard, unmodified surgical laparoscope and video system (EndoEye, Olympus Medical, Hamburg, Germany). This is the standard-of-care for these patients. During a standard procedure of upper lobectomy, segmental arteries are identified and ligated one at a time. Therefore, the investigators can create perfusion maps after ligation of the first segmental artery to identify the segment. The images will be shown to the surgeon postoperatively. The interlobar and intersegmental planes determined by PerfusiX-Imaging will be compared to the interlobar and intersegmental planes determined by ICG-Fluorescence imaging and the surgical eye.

5 TREATMENT OF SUBJECTS 5.1 Investigational product/treatment The investigational medical device is a medical imaging device that uses LSCI as a technology to image perfusion to identify the intersegmental planes. This technology is referred to in literature as laser speckle contrast imaging, laser speckle contrast analyses or laser speckle perfusion imaging. There is no change in treatment for the patients included in this study. The ICG-fluorescence device (Olympus, Hamburg, Germany) is a CE-certified device that is used on label.

5.2 Use over co-intervention (if applicable) Not applicable. 5.3 Escape medication (if applicable) Not applicable.

6 INVESTIGATIONAL DEVICE 6.1 Name and description of investigational medical device The investigational device is still in the development stage and only used for research purposes. The intraoperative imaging will be performed using a combination of our device and the OTV-S300 endoscopic video system (Olympus Surgical, Hamburg, Germany) with the EndoEye HD-II endoscope (Olympus Surgical, Hamburg, Germany).

6.1.1 Positioning in the operating room Positioning of the research set-up is outside the sterile zone of the operating room (OR). The fibreoptic cable between the white light source and the endoscope will be replaced by a connection between the white light source and the investigational medical device.

6.2 Summary of findings from non-clinical studies There is no literature on intersegmental plane detection using LSCI available. 6.3 Summary of findings from clinical studies There is no literature on intersegmental plane detection using LSCI available. 6.4 Summary of know and potential risks and benefits See IMDD (Version 1.1, November 2020, section 5) for a summary of known and potential risks and benefits of endoscopic LSCI.

7 NON-INVESTIGATIONAL PRODUCT 7.1 Name and description of non-investigation product(s) 7.1.1 Olympus surgical OTV-S300 video processor The OTV-S300 is an all-in-one 2D/3D processor and light source for endoscopic surgeries. It is capable of both 2D and 3D observation packed in a compact system for a simplified workflow. It has an LCD touch panel that allows for presets for easy preparation and maintenance. It has an LED light source which produces good natural colour reproduction with the combination of enhanced imaging processes. It has spectral light observation with narrowband imaging and two modes of IR-observation. A detailed description of the interface between PerfusiX-Imaging and the OTV-S300 can be found in the IMDD (Version 1.1, November 2020, section 1).

7.1.2 The EndoEye HD II videoscope delivers the innovative combination of distal-chip (chip-on-the-tip) and high-definition technology to provide surgeons with excellent images during endoscopic imaging. The HDII supports narrow band imaging. An advanced optical design provides greater depth of field, eliminating the need for manual focusing and other scope features include a digital zoom and fog-free heating function. The endoscope is fully autoclavable and the all-in-one design integrates the light cable and camera system into the endoscope for improved ergonomics and easier setup. A detailed description of the interface between PerfusiX-Imaging and the EndoEye HD II can be found in the IMDD (Version 1.1, November 2020, section 1) 7.1.3 Olympus ICG-fluorescence system The ICG-fluorescence system is produced by Olympus. The light source required for excitation of the ICG is the CLS-S200-IR that works in combination with the OTV-S300 video processor. The Olympus CH-S200 video head in combination with the Olympus IR telescope is the endoscope setup. This is the more traditional camera head - optics combination compared to the EndoEye. This system is installed in the MCL according to the ICG protocol found in attachment K6.16 7.2 Summary of findings from non-clinical studies Not applicable. 7.3 Summary of findings from clinical studies ICG-fluorescence imaging has been reported to determine the intersegmental planes. A recent study by Sun et al. has compared the inflation-deflation method and ICG-fluorescence imaging for the intersegmental plane determination in 19 patients13. Their results show that both methods were in total concordance with regards to the intersegmental demarcation. Other studies report larger patient groups. For example, Pischik et al. has assessed the safety and effectiveness of ICG-fluorescence imaging in 86 patients6. They were able to detect well defined fluorescence borders in 95.6% of the cases and had a fair explanation why the 4.4% failed. They concluded that ICG-fluorescence imaging is a safe and effective method for verification of anatomic segment borders. A feasibility study in 149 patients by Matsuura et al. also concluded that ICG-fluorescence is feasible and effective with a intersegmental line visible in a mere 98% of the patients14.

7.4 Summary of known and potential risks and benefits Not applicable. 7.5 Description and justification of route of administration and dosage See attachment K6.16 7.6 Dosages, dosage modifications and method of administration See attachment K6.16 7.7 Preparation and labelling of non-investigational medicinal product See attachment K6.16 7.8 Drug accountability Not applicable.

8 METHODS 8.1 Study parameters/endpoints 8.1.1 Study parameter/endpoint Due to the explorative character of this study, there is no formal hierarchy in the respective endpoints of this study. In this, all endpoints will add to the overall assessment of the feasibility of the PerfusiX-imaging derived visual feedback.

The investigators will look at the ability of PerfusiX-Imaging of detecting the interlobar and intersegmental planes.

In addition to this, the investigators will assess the conformity of the location of the interlobar and intersegmental planes as indicated by PerfusiX-imaging, compared to the location of the planes as indicated by the standard-of-care modalities, i.e., ICG-fluorescence imaging and the surgical eye.

The investigators will measure the time required for the capture of images with PerfusiX-Imaging to acquire the visual feedback for the surgeon.

To further assess the feasibility, the investigators will determine the cut-off values with the highest sensitivity and specificity with regards to the level of perfusion of lung tissue.

The interpretability of the visual feedback provided by PerfusiX-Imaging by the end-user will be assessed to get a sense of useability for the surgeon.

8.1.2 Other study parameters/endpoints (if applicable)

- Not applicable 8.2 Randomization, blinding and treatment allocation The current study is a non-randomized, non-blinded, prospective, single-centre in which all patients are scheduled to undergo a lobectomy according to standard care. There is no difference in therapeutic procedure among included patients.

8.3 Study procedures 8.3.1 Inclusion procedure Potential eligible patients are identified by their treating physician (in Dutch: hoofdbehandelaar). The treating physician will assess eligibility by checking in- and exclusion criteria based on the available data (according to paragraph 4.2 and 4.3). If a patient is found to be eligible to participate in the study, he or she will receive oral information about the study during a standard visit to the outpatient clinic, several days prior to surgical procedure. In addition, he or she will receive written study information (together with the standard information) from the medical assistant after the visit to the treating surgeon and is asked to consider participation. The patients will be informed about the aim of the study, the procedures and associated risks before enrolment into the study. Also, patients will be informed as to the strict confidentiality of their data.

Two weeks after receiving the information about the study, patients can inform their treating physician or the secretary staff of the Department of Surgery of theChirurgie MCL in person, by phone, mail or e-mail to confirm that they are willing to participate in this study. When patients agree to participate, signed written informed consent is obtained. For more specified information about informed consent, see chapter 11.2.

8.3.2 Image acquisition protocol The patient will be treated according to treatment plan as was established by the treating physician. The surgical procedure is executed as is deemed appropriate by the surgeon. The imaging acquisition protocol is executed on the to-be-excised lobe as described in Table 1. There will be two LSCI imaging moments during surgery. These imaging moment will be performed after ligation of the segmental vascularization, but before administration of ICG. This way, the recording is purely based on visual feedback from Laser Speckle Imaging, and there will be no bias based on the interpretation of ICG. The surgeon will not be able to see the LSCI images during the procedure. The LSCI researcher present in the OR will verbally guide the surgeon only with regards to positioning of the scope in order to acquire images that can be used to analyze. The researcher will not communicate any interpretation regarding position and deminsions of the plane. Depending on the procedure, a third measurement can be made in case an additional segment is isolated. Additionally, ICG-imaging will be performed. The imaging moments are (1) after ligating the first segmental arteries in the to-be-excised lobe, (2) after optional clipping of other segmental arteries in the to-be-excised lobe and (3) after ligation of all arteries of the to-be-excised lobe. The LSCI images will not be shown to the operating surgeon during surgery, but will be reviewed by the operating surgeon after the procedure has finished.

8.4 Withdrawal of individual subjects Subjects can leave the study at any time prior to surgery for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

8.4.1 Specific criteria for withdrawal (if applicable) Subjects will be withdrawn from the study when no surgery will be performed. 8.5 Replacement of individual subjects after withdrawal Patient who are withdrawn will be replaced in this study. 8.6 Follow-up of subjects withdrawn from treatment Not applicable. 8.7 Premature termination of the study 8.7.1 Termination based on safety aspects Not applicable 8.7.2 Termination based on other aspects The study will be suspended based on urgent medical or ethical considerations as decided by the principal investigators. In case of termination of the study, the institution, regulatory authorities, CCMO and the METC of the study centre will be informed.

9 SAFETY MONITORING 9.1 Temporary halt for reasons of subject safety In accordance to section 10, subsection 4 of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardize subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

9.2 AEs, SAEs 9.2.1 Adverse events (AEs) Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded.

9.2.2 Serious adverse events (SAEs) A serious adverse event is any untoward medical occurrence or effect that

* results in death;
* is life threatening (at the time of the event);
* requires hospitalization or prolongation of existing inpatients' hospitalization;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect; or
* any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator.

An elective hospital admission will not be considered as a serious adverse event.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within seven days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of eight days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

9.2.3 Suspected unexpected serious adverse reactions (SUSARs) Not applicable. 9.3 Annual safety report Not applicable. 9.4 Follow-up of adverse events All AEs that are related to the investigational medical product will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist. SAEs need to be reported till end of study within the Netherlands, as defined in the protocol.

9.5 Data Safety Monitoring Board (DSMB) An independent external Data Safety Monitoring Board of experts will not be instituted.

10 STATISTICAL ANALYSIS The overall aim of this study is to see if PerfusiX-Imaging can be used to determine the intersegmental planes.

10.1 Secondary study parameter(s) The total number of interlobar and intersegmental planes as detected using PerfusiX-Imaging that are in concordance with the interlobar and intersegmental planes as detected using ICG-fluorescence imaging and the surgical eye (descriptive statistics, percentage).

10.2 Other study parameters Not applicable. 10.3 Interim analysis (if applicable) Not applicable.

11 ETHICAL CONSIDERATIONS 11.1 Regulation statement The study will be conducted according to the principles of the Declaration of Helsinki (Fortaleza, Brazil, 2013 amendment) and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other guidelines, regulations and Acts. The protocol has been written and the study will be conducted according to the ICH Harmonized Tripartite Guideline for Good Clinical Practice. The protocol will be approved by the Local, Regional or National Ethics Committees.

11.2 Recruitment and consent Recruitment is done by the operating surgeon of the patient. All subjects are informed and asked for their consent. The minimal time between first appointment with doctor and surgery is 2 weeks, what results in a minimal time of 2 weeks for consideration.

Written informed consent must be obtained for all patients included in the study before they are registered in the study. Patients must be given adequate opportunity to read the information and enquire about details of the study before consent is given. This implies that the written informed consent form will be signed and personally dated by the patient. The informed consent statement will be signed and dated by the investigator afterwards and the patient will receive a copy. The general physician of each patient will be informed about the enrolment of the patient to the study.

11.3 Objection by minors or incapacitated subjects (if applicable) Not applicable. 11.4 Benefits and risk assessment, group relatedness All patients included in the study will be treated comparable with patients not included in the study. The difference between non-included and included patients is prolonged operating time. Prolonged operating time can increase the risk for patients, (e.g., infection (although this is rather minimal) and prolonged narcosis. The results do not immediately benefit the patients included in this study, but could help future patients to improve patient outcome.

11.5 Compensation for injury

The sponsor/investigator has a liability insurance which is in accordance with article 7 of the WMO. The sponsor (also) has insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO). This insurance provides cover for damage to research subjects through injury or death caused by the study. The total amounts of insurance are as follows:

1. A maximum of €650.000 (i.e. six hundred and fifty thousand euros) for death or injury for each subject who participates in this current research;
2. A maximum of €5.000.000 (i.e. five million five hundred thousand euros) for death or injury for all subjects who participate in this current research;
3. A maximum of €7.500.000 (i.e. seven million five hundred thousand euros) for the total damage that becomes apparent at the study participant in research which was conducted by the Medical Center Leeuwarden. Act in each year of insurance coverage.

The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

11.6 Incentives (if applicable) Not applicable. 12 ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION 12.1 Handling and storage of data and documents Data of patients will be handled confidentially and a coded identification number (study protocol number 'PORTION' followed by number of inclusion (for example PORTION01) will be used to link the data to the specific patient. Data that can be linked to a specific patient will be stored separately. The principal investigator safeguards the key to the code. The handling of the personal data complies with the EU General Data Protection Regulation and the Dutch Act on Implementation of the General Data Protection Regulation (in Dutch: Uitvoeringswet AVG, UAVG)). These data will be stored at the specific site for at least fifteen years. For software adjustments a software engineer from ZiuZ Research BV can have access to only the images.

12.2 Monitoring and Quality Assurance Not applicable. 12.3 Amendments

Amendments are changes made to the research after a favourable opinion by the accredited METC has been given. All amendments will be notified to the METC that gave a favourable opinion. A 'substantial amendment' is defined as an amendment to the terms of the METC application, or to the protocol or any other supporting documentation, that is likely to affect to a significant degree:

* the safety or physical or mental integrity of the subjects of the trial;
* the scientific value of the trial;
* the conduct or management of the trial; or
* the quality or safety of any intervention used in the trial. All substantial amendments will be notified to the METC and to the competent authority. Non-substantial amendments will not be notified to the accredited METC and the competent authority, but will be recorded and filed by the sponsor.

12.4 Annual progress report The sponsor/investigator will submit a summary of the progress of the trial to the accredited METC once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

12.5 Temporary halt and (prematurely) end of study report The investigator/sponsor will notify the accredited METC of the end of the study within a period of 8 weeks. The end of the study is defined as the last patient's last visit. The sponsor will notify the METC immediately of a temporary halt of the study, including the reason of such an action. In case the study is ended prematurely, the sponsor will notify the accredited METC within 15 days, including the reasons for the premature termination. Within one year after the end of the study, the investigator/sponsor will submit a final study report with the results of the study, including any publications/abstracts of the study, to the accredited METC.

12.6 Public disclosure and publication policy The financial sponsor of the study is LIMIS Development BV (Principal Investigator dr. E.C. Boerma). There are no restrictions towards publication; the study is registered in a public trial registry (clinicaltrials.gov) and with the CCMO number NL82338.099.22.

13 STRUCTURED RISK ANALYSIS 13.1 Potential issues of concern

1. Level of knowledge about mechanism of action NA
2. Previous exposure of human beings with the test product(s) and/or products with a similar biological mechanism NA
3. Can the primary or secondary mechanism be induced in animals and/or in ex-vivo human cell material? NA
4. Selectivity of the mechanism to target tissue in animals and/or human beings NA
5. Analysis of potential effect NA
6. Pharmacokinetic considerations NA
7. Study population NA
8. Interaction with other products NA
9. Predictability of effect NA
10. Can effects be managed? NA

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo upper left or right lobectomy
* Age 18 years or older
* Written informed consent

Exclusion Criteria:

- Medical or psychiatric conditions that compromise the patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients meeting the eligibility criteria and scheduled to undergo a lobectomy in the Medical Centre Leeuwarden
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The ability of PerfusiX-Imaging of detecting the interlobar and intersegmental planes. | 1 day
  - The total number of interlobar and intersegmental planes detected using PerfusiX-Imaging (yes/no, percentages, 95% Confidence Interval).
The ability of PerfusiX-Imaging of detecting the interlobar and intersegmental planes compared to ICG and surgical eye | 1 day
  - Comparison between total amount of detected planes using PerfusiX-Imaging, ICG and the surgical eye (yes/no per modality, percentages, 95% Confidence Interval).
Assessing the conformity of plane location between PerfusiX-Imaging and ICG-fluorescence/surgical eye. | 1 day
  - Difference in location of planes of LSCI, compared to ICG and the surgical eye (means with standard deviation, median with range)
Required time to capture images with PerfusiX-Imaging | 1 day
  - Time per measurement and total time per procedure in minutes (means with standard deviation, median with range)
Interpretability of visual feedback derived from PerfusiX-Imaging by the operating surgeon. | 1 day
  - Overlap in surface between modalities (means with standard deviation, median with range)
Determination of Laser Speckle Perfusion Unit (LSPU) cut-off value with the highest sensitivity and specificity | during the total inclusion time, depending on the time needed to include all required patients.
  - ROC curve analysis (Laser Speckle values referenced to standard care (ICG)) and anatomical feature (interlobar fissure).

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andolfi M, Potenza R, Seguin-Givelet A, Gossot D. Identification of the intersegmental plane during thoracoscopic segmentectomy: state of the art. Interact Cardiovasc Thorac Surg. 2020 Mar 1;30(3):329-336. doi: 10.1093/icvts/ivz278. PMID 31773135
- [Background] Funai K, Kawase A, Shimizu K, Sekihara K, Yamashita T, Shiiya N. Fluorescence navigation with indocyanine green for identification of intersegmental planes using a photodynamic eye camera. J Thorac Dis. 2020 Sep;12(9):4817-4824. doi: 10.21037/jtd-20-1448. PMID 33145054
- [Background] Zhang Z, Liao Y, Ai B, Liu C. Methylene blue staining: a new technique for identifying intersegmental planes in anatomic segmentectomy. Ann Thorac Surg. 2015 Jan;99(1):238-42. doi: 10.1016/j.athoracsur.2014.07.071. Epub 2014 Nov 14. PMID 25440279
- [Background] Nex G, Schiavone M, De Palma A, Quercia R, Brascia D, De Iaco G, Signore F, Panza T, Marulli G. How to identify intersegmental planes in performing sublobar anatomical resections. J Thorac Dis. 2020 Jun;12(6):3369-3375. doi: 10.21037/jtd.2020.01.09. PMID 32642262
- [Background] Oh S, Suzuki K, Miyasaka Y, Matsunaga T, Tsushima Y, Takamochi K. New technique for lung segmentectomy using indocyanine green injection. Ann Thorac Surg. 2013 Jun;95(6):2188-90. doi: 10.1016/j.athoracsur.2012.12.068. PMID 23706452
- [Background] Pischik VG, Kovalenko A. The role of indocyanine green fluorescence for intersegmental plane identification during video-assisted thoracoscopic surgery segmentectomies. J Thorac Dis. 2018 Nov;10(Suppl 31):S3704-S3711. doi: 10.21037/jtd.2018.04.84. PMID 30505555
- [Background] Briers JD, Fercher AF. Retinal blood-flow visualization by means of laser speckle photography. Invest Ophthalmol Vis Sci. 1982 Feb;22(2):255-9. PMID 7056639
- [Background] Draijer M, Hondebrink E, van Leeuwen T, Steenbergen W. Review of laser speckle contrast techniques for visualizing tissue perfusion. Lasers Med Sci. 2009 Jul;24(4):639-51. doi: 10.1007/s10103-008-0626-3. Epub 2008 Dec 3. PMID 19050826
- [Background] Boas DA, Dunn AK. Laser speckle contrast imaging in biomedical optics. J Biomed Opt. 2010 Jan-Feb;15(1):011109. doi: 10.1117/1.3285504. PMID 20210435
- [Background] Heeman W, Dijkstra K, Hoff C, Koopal S, Pierie JP, Bouma H, Boerma EC. Application of laser speckle contrast imaging in laparoscopic surgery. Biomed Opt Express. 2019 Mar 25;10(4):2010-2019. doi: 10.1364/BOE.10.002010. eCollection 2019 Apr 1. PMID 31086715
- [Background] Sun Y, Zhang Q, Wang Z, Shao F, Yang R. Is the near-infrared fluorescence imaging with intravenous indocyanine green method for identifying the intersegmental plane concordant with the modified inflation-deflation method in lung segmentectomy? Thorac Cancer. 2019 Oct;10(10):2013-2021. doi: 10.1111/1759-7714.13192. Epub 2019 Sep 3. PMID 31482671
- [Background] Matsuura Y, Mun M, Ichinose J, Nakao M, Nakagawa K, Okumura S. Recent fluorescence-based optical imaging for video-assisted thoracoscopic surgery segmentectomy. Ann Transl Med. 2019 Jan;7(2):32. doi: 10.21037/atm.2019.01.23. PMID 30854385